CLINICAL TRIAL: NCT04587973
Title: The Effectiveness of Bilateral Erector Spinae Plane Block (ESPB) in Laparoscopic Cholecystectomies. A Randomized, Controlled, Double Blind, Prospective, Trial
Brief Title: Bilateral Erector Spinae Plane Block (ESPB) in Laparoscopic Cholecystectomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Professor of Anesthesiology, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ESPB-Frida
Record Dates: First submitted 2020-10-08; First posted 2020-10-14 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Pain, Postoperative; Pain Syndrome; Pain, Acute; Anesthesia; Cholecystectomy; Erector Spinae Plane Block
MeSH Terms: conditions — Pain, Postoperative; Somatoform Disorders; Acute Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Dexmedetomidine (Active Comparator): Ropivacaine plus dexmedetomidine group - Preoperative bilateral erector spinae plane block with ropivacaine 0,375% (40 ml) plus dexmedetomidine 1 mcg/kg
  Interventions: Procedure: Group Dexmedetomidine
- Group Ropivacaine (Active Comparator): Plain ropivacaine group - Preoperative bilateral erector spinae plane block with ropivacaine 0,375% (40 ml)
  Interventions: Procedure: Group Ropivacaine
- Group Control (Placebo Comparator): Control group - Preoperative bilateral erector spinae plane block with N/S 0,9% (40 ml)
  Interventions: Procedure: Group Control

INTERVENTIONS:
Procedure: Group Dexmedetomidine — Ropivacaine plus dexmedetomidine group
  Arms: Group Dexmedetomidine
Procedure: Group Ropivacaine — Plain ropivacaine group
  Arms: Group Ropivacaine
Procedure: Group Control — Control group
  Arms: Group Control

SUMMARY:
The aim of the trial is to study the efficacy of bilateral Erector Spinae Plane Block (ESPB) in managing perioperative pain in patients who undergo elective laparoscopic cholecystectomy

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is one of the most common performed procedures of general surgery. Although it is performed with minimally invasive techniques, postoperative pain can be moderate to severe, requiring administration of large doses of opioids perioperatively in combination with other categories of analgesics in order to be relieved. Modern anesthesiology practices tend to limit the opioids administered to patients due to a variety of complications observed, specifically in certain populations (obese, elderly) and also due to the opioid crisis appearance in United States and in many European countries. As such, multimodal analgesia and opioid limitation is the cornerstone of modern perioperative pain management.

Peripheral nerve blocks and especially trunk blocks can play a significant role when confronting perioperative pain. Erector spinae Plane Block (ESPB) is a novel trunk block first described in order to relieve thoracic neuropathic pain. Since then, it was performed by anesthesiologists for chronic pain, acute post traumatic pain and in a wide variety of surgical procedures for postoperative analgesia.

There are no trials that study the efficacy of adding dexmedetomidine as an adjuvant to the local anesthetic in order to ameliorate the quality and extend the duration of the Erector Spinae Plane Block.

This trial is a randomized, controlled, double - blind, prospective trial, aiming at assessing the efficacy of bilateral Erector Spinae Plane Block (ESPB) in managing perioperative pain in patients who undergo elective laparoscopic cholecystectomy. In this trial, 60 patients (men and women), aged 18 to 70 years old that will undergo laparoscopic cholecystectomy which will be performed by the same experienced, surgical team, will be recruited.

Patients will be randomized into three groups, Group D (Ropivacaine plus dexmedetomidine group), Group R (Plain Ropivacaine group) and Group C (Control group).

The solutions that will be administered during the performance of ESPB, will be prepared by an independent anesthesiologist. The ultrasound image during the performance of ESPB, as well as the complications that may arise after the performance of the block, will be recorded.

The age, sex, American Society of Anesthesiologists (ASA) classification, height and weight of the participants, will be recorded.

After the induction of general anesthesia [propofol (2-3 mg/kg), fentanyl (2-3 γ/kg), rocuronium (0,6 mg/kg)], general anesthesia will be maintained with desflurane titration. In all patients, remifentanil infusion will be titrated in order to achieve intraoperative analgesia (Systolic Arterial Blood Pressure within the 20% of Baseline Systolic Blood Pressure). In all patients Paracetamol 1000 mg and Tramadol 100 mg will be administered, 30 minutes before the end of surgery. During surgery, vital signs, remifentanil infusion or other drugs that will be administered, will be recorded. At the end of surgery, Train of Four stimulation will be performed and in the presence of remaining neuromuscular blockade, sugammadex will be administered in the proper doses.

In all patients, post - operative analgesia will be offered with a Patient controlled Analgesia (PCA) pump, containing morphine. Lock - out period will be 10 minutes and the morphine dose will be 20 mcg/kg, without continuous infusion.

The duration of stay of the patient in Post Anesthesia Care Unit (PACU), will be recorded as well as the Aldrete Score and the vital signs the moment the patient leaves the PACU.

Postoperative pain will be recorded at arrival and discharge of the patient from the PACU, as well as 3, 6, 12 and 24 hours after the end of surgery, according to NRS pain scale. All patients will receive Paracetamol 1000 mg x 3 (iv) at the surgical ward.

Post - operative nausea and vomiting, morphine consumption and the vital signs of the patients will be recorded 3, 6, 12and 24 hours after surgery. The mobilization time, hospitalization time, as well as the satisfaction score of the patient in a scale from 1 to 6, 24 hours after the end of surgery will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II
* Laparoscopic cholecystectomy
* Elective surgery

Exclusion Criteria:

* Patient refusal
* Coagulation disorders
* Known allergies to local anesthetics
* Other contraindications to regional anesthesia
* Infection or anatomic anomalies on injection site
* Uncontrolled hypertension
* Severe liver or kidney disease
* Pregnancy
* Known depression or psychiatric disorders, dementia
* Drug or alcohol abuse
* Inadequate command of Greek language

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
pain score 3 hours postoperatively | 3 hours after surgery
  pain score by the use of Numeric Rating Scale (NRS) 3 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 6 hours postoperatively | 6 hours after surgery
  pain score by the use of Numeric Rating Scale (NRS) 6 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 12 hours postoperatively | 12 hours after surgery
  pain score by the use of Numeric Rating Scale (NRS) 12 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 24 hours postoperatively | 24 hours after surgery
  pain score by the use of Numeric Rating Scale (NRS) 24 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score on arrival to Post-Anesthesia Care Unit (PACU) | immediately postoperatively
  pain score by the use of Numeric Rating Scale (NRS) on arrival to PACU, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score at discharge from Post-Anesthesia Care Unit (PACU), ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable" | immediately postoperatively
  pain score by the use of Numeric Rating Scale (NRS) at discharge from PACU

SECONDARY OUTCOMES:
morphine consumption | 24 hours postoperatively
  morphine consumption through patient-controlled analgesia device for 24 hours postoperatively
satisfaction from postoperative analgesia | 24 hours postoperatively
  satisfaction from postoperative analgesia on a six-point Likert scale with 1 marked as minimal satisfaction and 6 as maximal satisfaction
mobilization time | 24 hours postoperatively
  time at which the patient mobilizes after surgery
hospitalization time | 72 hours postoperatively
  duration of hospital stay after surgery in days
intraoperative dose of remifentanil infusion (μg kg-1) | intraoperatively
  dose of required remifentanil intraoperatively to maintain systolic arterial blood pressure within the 20% of baseline value
Erector Spinae Plane Block-related complications | 48 hours postoperatively
  block-related complications at the site of the local anesthetic injection
Post Anesthesia Care Unit (PACU) duration of stay | immediately postoperatively
  duration of patient stay at PACU

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, PhD, DESA, Study Chair — Aretaieion University Hospital
Locations (1):
- George Papanikolaou, General Hospital of Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ibrahim M. Erector Spinae Plane Block in Laparoscopic Cholecystectomy, Is There a Difference? A Randomized Controlled Trial. Anesth Essays Res. 2020 Jan-Mar;14(1):119-126. doi: 10.4103/aer.AER_144_19. Epub 2020 Feb 3. PMID 32843804
- [Background] Herman JA, Urits I, Kaye AD, Urman RD, Viswanath O. Erector Spinae Plane Block (ESPB) or Quadratus Lumborum Block (QLB-II) for laparoscopic cholecystectomy: Impact on postoperative analgesia. J Clin Anesth. 2020 Nov;66:109958. doi: 10.1016/j.jclinane.2020.109958. Epub 2020 Jun 17. No abstract available. PMID 32563073
- [Background] Kwon HM, Kim DH, Jeong SM, Choi KT, Park S, Kwon HJ, Lee JH. Does Erector Spinae Plane Block Have a Visceral Analgesic Effect?: A Randomized Controlled Trial. Sci Rep. 2020 May 21;10(1):8389. doi: 10.1038/s41598-020-65172-0. PMID 32439926
- [Background] Peker K, Akcaboy ZN, Aydin G, Gencay I, Sahin AT, Kocak YF, Peker SA. The Effect of Erector Spinae Plane Block on Laparoscopic Cholecystectomy Anesthesia: Analysis of Opioid Consumption, Sevoflurane Consumption, and Cost. J Laparoendosc Adv Surg Tech A. 2020 Jul;30(7):725-729. doi: 10.1089/lap.2019.0809. Epub 2020 Feb 5. PMID 32023174
- [Background] Aygun H, Kavrut Ozturk N, Pamukcu AS, Inal A, Kiziloglu I, Thomas DT, Tulgar S, Nart A. Comparison of ultrasound guided Erector Spinae Plane Block and quadratus lumborum block for postoperative analgesia in laparoscopic cholecystectomy patients; a prospective randomized study. J Clin Anesth. 2020 Jun;62:109696. doi: 10.1016/j.jclinane.2019.109696. Epub 2019 Dec 18. PMID 31862217
- [Background] Raft J, Chin KJ, Gobert Q, Richebe P, Brulotte V. Defining the optimal analgesic strategy for erector spinae plane (ESP) blocks in unanticipated open cholecystectomy. Korean J Anesthesiol. 2019 Oct;72(5):504-505. doi: 10.4097/kja.d.18.00350. Epub 2018 Dec 28. No abstract available. PMID 30590914
- [Derived] Sifaki F, Mantzoros I, Koraki E, Bagntasarian S, Christidis P, Theodoraki K. The Effect of Ultrasound-guided Bilateral Erector Spinae Plane Block With and Without Dexmedetomidine on Intraoperative and Postoperative Pain in Laparoscopic Cholecystectomies: A Randomized, Controlled, Double-blind, Prospective Trial. Pain Physician. 2022 Oct;25(7):E999-E1008. PMID 36288585